CLINICAL TRIAL: NCT04741139
Title: Reduction of Adverse Events and Re-Presentation to Medical Care After Intravenous Immunoglobulin Treatment in Children With Immune Thrombocytopenia With a Scheduled Post-Infusion Medication Strategy
Brief Title: Post IVIG Medication in Children With Immune Thrombocytopenia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Megan Gilbert, Principal Investigator, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-47160
Record Dates: First submitted 2020-10-13; First posted 2021-02-05 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Single hospital system, single-arm year-long pilot to evaluate the feasibility of enrolling children with ITP who are receiving IVIG for treatment of disease to a scheduled post-infusion medication for 72 hours following IVIG infusion.
  This year-long feasibility pilot will test the (1) feasibility of enrollment and the willingness of families to participate in a scheduled medication regimen and (2) adherence of patients and families to the scheduled medication regimen. Clinical outcomes, as defined by rates of headache or nausea/vomiting or other adverse event following IVIG, return to medical care, and need for further laboratory or imaging studies, will be collected. These rates will be compared to retrospective, historical data from Texas Children's Hematology Center from 2010 to 2019. However, due to the rate at which these events occur following IVIG, this feasibility pilot is not fully powered to detect differences in clinical outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Scheduled post-IVIG medication (Experimental): Utilization of post-IVIG medication with acetaminophen and diphenhydramine on a scheduled basis of 72 hours post-infusion.
  Interventions: Drug: Acetaminophen and Diphenhydramine Only Product

INTERVENTIONS:
Drug: Acetaminophen and Diphenhydramine Only Product — Using a scheduled medication regimen of diphenhydramine and acetaminophen following IVIG medication to evaluate feasibility of enrollment, medication adherence, side effects related to study medication and IVIG.

SUMMARY:
This study is a single hospital system, single-arm year-long pilot to evaluate the feasibility of enrolling children with ITP who are receiving IVIG for treatment of disease to a scheduled post-infusion medication for 72 hours following IVIG infusion.

This year-long feasibility pilot will test the (1) feasibility of enrollment and the willingness of families to participate in a scheduled medication regimen and (2) adherence of patients and families to the scheduled medication regimen. Clinical outcomes, as defined by rates of headache or nausea/vomiting or other adverse event following IVIG, return to medical care, and need for further laboratory or imaging studies, will be collected. These rates will be compared to retrospective, historical data from Texas Children's Hematology Center from 2010 to 2019. However, due to the rate at which these events occur following IVIG, this feasibility pilot is not fully powered to detect differences in clinical outcomes.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is the most common acquired immune cytopenia in childhood, affecting 4-6 in 100,000 children. The pathophysiology of ITP is highly complex and incompletely understood. Accepted mechanisms include immune dysregulation caused by an often unidentified trigger leading to the formation of anti-platelet antibodies and antibody-mediated reticuloendothelial clearance. Cell-mediated platelet destruction and disruption of T cell homeostasis are also well described. ITP is also characterized by impaired platelet production due to antibody effect in the bone marrow and subsequent megakaryocyte ultrastructural abnormalities.

Children with ITP generally present with a sudden onset of symptoms. Bleeding tendency is variable, but the vast majority of children will experience cutaneous bleeding symptoms including bruising and petechiae. More extensive bleeding ranging from extensive oral bleeding, gastrointestinal bleeding, menorrhagia, or other significant bleeding necessitating urgent medical intervention develops in up to 20% of patients.8 Intracranial hemorrhage (ICH), the most feared and devastating complication of ITP, occurs in approximately 0.5% of pediatric patients. Bleeding phenotype is unable to be reliably predicted at diagnosis. In children who present with mucosal or more significant bleeding, treatment is indicated to achieve rapid hemostasis by increase in platelet count. Intravenous immunoglobulin (IVIG) is a commonly utilized first line agent to reduce bleeding symptoms and improve the platelet count to a hemostatic range within 24-48 hours of administration. The mechanism of action of IVIG in ITP is currently incompletely understood and likely involves multiple immunomodulatory mechanisms. Previous data has suggested IVIG leads to a rise in platelet count via blockade of Fc receptors on phagocytic cells within the reticuloendothelial system. Another hypothesis suggests IVIG upregulates the expression of the inhibitory IgG Fc receptor 2B encoded by FCGR2B gene, thus leading to decreased cell mediated destruction and decreased anti-platelet antibody production.14 Following IVIG administration, an improvement in clinical bleeding and an associated rise in platelet count is seen in approximately 75% of children with ITP

IVIG is a polyclonal antibody preparation developed from pooled donor plasma from 15,000 to 60,000 donors depending on the preparation utilized. The safety and efficacy of IVIG in patients with ITP has been demonstrated in multiple clinical trials, and IVIG is considered a first line therapy for the treatment of children with ITP. Overall, IVIG is well tolerated across patients with a spectrum of diseases. The majority of reported adverse events are mild, transient, and infusion related. The most commonly reported immediate adverse events include headache, fever, nausea/vomiting, malaise, back pain, flushing, and chills. In comparison to other patient populations who receive IVIG, patients with ITP carry the unique risk for intracranial hemorrhage due to profound thrombocytopenia. Mild side effects such as headache and nausea/vomiting can easily be attributed to recent IVIG administration in non-thrombocytopenic populations. However, these symptoms overlap with the heralding symptoms of an intracranial hemorrhage which, due to high morbidity and mortality, must not go undiagnosed in patients with ITP. To decrease the percentage of patients experiencing these immediate, infusion associated symptoms, patients with ITP at most pediatric centers are routinely pre-medicated with a single dose of acetaminophen and diphenhydramine prior to IVIG infusion.21 However, post-infusion medication regimens differ amongst providers and pediatric centers and frequently utilized acetaminophen and diphenhydramine as these symptoms arise.

Peak IgG concentration following IVIG administration occurs in the cerebrospinal fluid (CSF) between 24-48 hours after infusion. The common events of headache, nausea, and vomiting often peak during this time, when most patients have already been discharged from medical care. Headache and associated nausea/vomiting are particularly worrisome in patients with ITP given the risk for ICH and overlap of symptoms at presentation. Aseptic meningitis, a rare and serious adverse event following IVIG infusion, presents with headache, nausea/vomiting, nuchal rigidity, and fever. The development of aseptic meningitis is hypothesized to be dose dependent and has been noted to cluster within patients who suffer from migraines.

At Texas Children's Hospital, most children prescribed IVIG receive Gamunex-C, which has a reported incidence of headache in 30-50% of patients. At the onset of symptoms, patients typically remain severely thrombocytopenic and at highest risk of ICH. Many of these patients will develop symptoms severe enough to necessitate return to medical care, additional laboratory studies, and computed tomography (CT) of the head to rule out ICH. Texas Children's Hematology Center data reveals 28% of the 473 IVIG infusions administered to patients for ITP between 2010 and 2016 resulted in the report of headache or nausea/vomiting. Seventy-seven percent (103/133) of these infusions resulted in the patient developing symptoms sufficiently severe to cause re-evaluation by a medical provider. Subsequent urgent visits often come at significant expense. Of the 133 infusions resulting in the report of headache and/or nausea/vomiting, 45% (60/133) required additional lab work and 27% (36/133) required imaging via CT to rule out ICH ( please see Figure 1 in the full protocol). These 36 patients who required urgent head CTs represent 7.6% of all IVIG infusions administered for ITP between 2010 and 2016 (American Society of Hematology Conference Abstract 2018; further cohort data analysis in process).

The etiology of these neurologic IVIG-associated adverse events is not well understood. It is currently hypothesized that central nervous system (CNS) symptoms ranging from headache to aseptic meningitis following IVIG administration may represent a spectrum of symptoms secondary to IgG-mediated meningeal inflammation. This hypothesis is based off cerebrospinal fluid (CSF) analysis in patients who developed aseptic meningitis following IVIG. CSF demonstrated the presence of allogeneic IgG as well as pleocytosis with neutrophil predominance. As the pathophysiology underlying the development of these adverse events is currently not fully understood, it is reasonable to trial the safe pediatric medications that are already employed in premedication regimens. It is for this reason the investigators propose the use of acetaminophen and diphenhydramine for the post-IVIG infusion medication regimen.

Currently, no evidence-based guideline exists for the administration of prophylactic medications following IVIG infusions as these specific IVIG side effects are of less concern in non-thrombocytopenic patients. The 2011 American Society of Hematology ITP Clinical Practice Guidelines found insufficient evidence to recommend or oppose routine premedication prior to IVIG. The newly released 2019 Guidelines note that headache can be particularly problematic, however they do not recommend a specific avoidance strategy. While providers often pre-medicate, post-infusion medication practices are entirely physician dependent and frequently involve the use of acetaminophen and diphenhydramine as symptoms arise. The investigators hypothesize that an alternative approach to post-infusion practices may alter IVIG-related symptomatology, particularly those symptoms most alarming in a patient with thrombocytopenia and at risk for ICH. Scheduled post-infusion medication with acetaminophen and diphenhydramine may decrease the rate of worrisome symptoms in patients with ITP and subsequently decrease the need to return to medical care where additional laboratory and imaging studies are often performed to further assess for ICH. The ability of routine post-infusion medication to decrease the rate of adverse events and subsequent return to medical care has yet to be studied in patients with ITP.

It is unknown whether families of children with ITP are willing to enroll in a clinical trial to evaluate the effects and potential benefits of scheduled post-infusion. Additionally, it is unknown to what degree adherence to scheduled post-infusion medication can be achieved. In order to determine if enrollment and adherence can be achieved, the investigators plan to conduct a year-long feasibility study in patients in whom IVIG is indicated for treatment of bleeding symptoms and/or risk associated with ITP (Figure 2). The results of this feasibility study will assess the ability to successfully conduct future comparative randomized control trials (RCTs). This single-arm feasibility study with comparison to Texas Children's Hematology Center historical data will also provide preliminary clinical data regarding rates of return to medical care and additional medical interventions. Further RCTs will be critical to determine if the number of patients who must return to care and undergo further testing can be decreased with a scheduled post-infusion medication regimen. These data will inform future clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ITP confirmed by hematology team.
* Patient receiving IVIG for a clinical indication as determined by primary hematologist. IVIG can be administered in the inpatient, outpatient, and emergency room settings.
* Age 0 to 18 years

Exclusion Criteria:

* Patients with a history of anaphylaxis to IVIG infusion.
* Patients receiving IVIG for indications other than ITP.
* Patients who have previously received IVIG or who receive multiple IVIG infusions within the study period.
* Patients who require additional platelet direct therapies including corticosteroids, anti-D immunoglobulin, rituximab, or thrombopoietin receptor agonists.
* Other cause of thrombocytopenia (congenital thrombocytopenias, drug induced thrombocytopenia, bone marrow failure, liver disease, etc.) apparent by history and physical examination, and/or laboratory tests.
* Inability to tolerate oral medications
* Other medical or social factors at discretion of treating physician such as ability to follow-up, etc.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Eligible Patients Agreeing to Enrollment | 12 months
  Patients who are considered eligible for study participation and are approached by the research team to participate will be included in the determination of enrollment feasibility.

SECONDARY OUTCOMES:
Percentage of Enrolled Patients who Achieve Medication Adherence | 12 months
  Patients and families will be considered adherent to the medication regimen if >75% of the scheduled doses are administered (average of 3 of 4 daily doses given). A patient must meet the following two criteria to be considered adherent:
  1. The patient received on average at least 75% of the scheduled doses across the 72 hours study period
  2. The patient received at least 75% of the doses scheduled to be given within the first 24 hours of the study period
Rate of Return to Medical Care for Emergent Evaluation | 72 hours following IVIG for each patient
  The rate of return to medical care for emergent evaluation, along with additional clinical outcomes as detailed in outcomes 4-6, will be collected. This rate will be compared to retrospective, historical data from Texas Children's Hematology Center from 2010 to 2019. However, due to the rate at which these events occur following IVIG, this feasibility pilot is not fully powered to detect differences in clinical outcomes. This data will provide important preliminary clinical data regarding rates of return to medical care and additional medical interventions.
Rates of IVIG-Associated Adverse Drug Events | 72 hours following IVIG for each patient
  The rates of headache, nausea/vomiting, and other patient reported adverse event following IVIG will be collected. These rates will be compared to retrospective, historical data from Texas Children's Hematology Center from 2010 to 2019. However, due to the rate at which these events occur following IVIG, this feasibility pilot is not fully powered to detect differences in clinical outcomes. This data will provide important preliminary clinical data regarding rates of return to medical care and additional medical interventions.
Rate of Laboratory Evaluation with Platelet Count During Emergent Medical Evaluation | 72 hours following IVIG for each patient
  In addition to the rate at which patients return to medical care for emergent evaluation after IVIG, the rate of subsequent laboratory evaluation, specifically platelet count, will be collected. This rate will be compared to retrospective, historical data from Texas Children's Hematology Center from 2010 to 2019. However, due to the rate at which these events occur following IVIG, this feasibility pilot is not fully powered to detect differences in clinical outcomes. This data will provide important preliminary clinical data regarding rates of return to medical care and additional medical interventions.
Rate of Patients Requiring Head CT During Emergent Medical Evaluation | 72 hours following IVIG for each patient
  The rate of patients who require CT of the head during return to medical care for emergent evaluation will be collected. This rate will be compared to retrospective, historical data from Texas Children's Hematology Center from 2010 to 2019. However, due to the rate at which these events occur following IVIG, this feasibility pilot is not fully powered to detect differences in clinical outcomes. This data will provide important preliminary clinical data regarding rates of return to medical care and additional medical interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States